CLINICAL TRIAL: NCT00536016
Title: A Phase 1 Open Label Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of Single and Repeated Doses of JSM6427 Following Administration by Intravitreal Injection in Patients With Neovascular AMD
Brief Title: A Phase 1 Safety Study of Single and Repeated Doses of JSM6427 (Intravitreal Injection) to Treat AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jerini Ophthalmic (Industry)
Responsible Party: Jerini Ophthalmic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JO642701
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Macular Degeneration
Keywords: AMD; Neovascular Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — JSM6427

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: JSM6427 — Weekly intravitreal injections for up to 4 weeks, first dose strength is one dose below the MTD. Dose strength concentrations: 1.5 mg/ml, 3 mg/ml, 7.5 mg/ml 04 15 mg/ml.

SUMMARY:
The purpose of this study is to determine the way and rate that the study medication, JSM6427 a potent, highly specific integrin α5β1-antagonist is absorbed, broken-down and eliminated from the body when it is given as a single dosage strength by injection into the eye. Repeated dosages will also be given to determine the highest safe dose.

DETAILED DESCRIPTION:
In non-clinical models, JSM6427 can lead to the inhibition and regression of choroidal neovascularization, making α5β1 an attractive target for therapeutic strategies directed at pathological angiogenesis. JSM6427 may also interfere with other key processes in the pathogenesis of AMD, namely inflammation and fibrosis. Further, non-clinical data show that JSM6427 inhibits scarring and inflammation. Thus, JSM6427 may target multiple important pathways in the pathogenesis of neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity in the study eye between 5 and 7 letters inclusive using and ETDRS chart (Snellen equivalent of appx. 20/800 to 20/40.
* Subfoveal choroidal neovascularization (CNV) due to AMD.
* Total area of the lesion (including blood, neovascularization and scar/atrophy) must be ≤ 12 DA, of which at least 25% must be active CNV.
* For patients with occult or non classic CNV; there must be the presence of subretinal hemorrhage (but still comprising no more than 50% of the lesion) and/or documented evidence of three or more lines of vision loss (ETDRS or equivalent) during the previous 12 weeks.
* Clear ocular media and adequate pupillary dilatation to permit good stereo fundus photography for screening.
* Intraocular pressure of 21 mm Hg or less.
* Retinal thickness ≥ 250 μm by OCT.
* Normal screening ERG
* Normal ECG

Exclusion Criteria:

* PDT within 120 days prior to screening in the study eye.
* Previous therapeutic radiation to the eye.
* Any retinovascular disease or retinal degeneration other than AMD.
* Serous pigment epithelial detachment without the presence of neovascularization.
* Presence of pigment epithelial tears or rips.
* Previous posterior vitrectomy or retinal surgery.
* Any periocular infection in the past 4 weeks.
* Concomitant therapy with anti-VEGF therapies, e.g. Avastin, Lucentis or Macugen, or previous use of these agents within 60 days of screening in the study eye.
* Concomitant therapy with intravenous or intravitreous corticosteroids or use within 90 days of screening.
* Cataract surgery in the study eye within three months of screening.
* Intraocular surgery in the study eye within three months of screening.
* Presence of ocular infection in the study eye.
* Presence of severe myopia (-8 diopters or greater) in the study eye.
* Allergy to or prior significant adverse reaction to fluorescein.
* Any major surgical procedure within one month of trial entry.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability to determine the MTD | 2 weeks after each dose

SECONDARY OUTCOMES:
To evaluate the systemic pharmacokinetics of JSM6427 following single and repeat doses by intravitreal injection and to assess exploratory efficacy potential of JSM6427 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Adamis, MD, Study Chair — Jerini Ophthalmic
Locations (9):
- United States (9):
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - William Beaumont Research Institute, Royal Oak, Michigan
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Research Institute of Texas, Abilene, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - Valley Retina Institute, McAllen, Texas